CLINICAL TRIAL: NCT04570111
Title: A Modern Approach to Dietary Management of Gestational Diabetes Mellitus
Brief Title: MOD Diet in Gestational Diabetes Mellitus
Acronym: MOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate number of eligible participants
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 145905
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Gestational Diabetes
Keywords: diet therapy; patient education
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Diet (Active Comparator): After the controlled feeding study, participants in this group will follow the standard care diet for the remainder of pregnancy with the assistance of a study dietitian. The standard care study diet will provide the standard 40% Carb/20% Pro/40% Fat as energy, distributed consistently across 3 meals and 2 snacks.
  Interventions: Other: Standard Care Diet
- Macro-Optimized Diet (MOD) (Experimental): After the controlled feeding study, participants in this group will follow the MOD diet for the remainder of pregnancy with the assistance of a study dietitian. The MOD diet will differ from control by macronutrient distribution at breakfast specifically, but also at each eating occasion, although the daily macronutrient distribution is equal to the control diet. At breakfast, the MOD diet will provide 10% Carb/30% Pro/60% Fat.
  Interventions: Other: MOD Diet

INTERVENTIONS:
Other: MOD Diet — The macro-optimized diet alters the timing of macronutrient intake to provide fewer carbohydrates at breakfast, while maintaining recommended amounts of macronutrients delivered throughout the course of the day
  Arms: Macro-Optimized Diet (MOD)
Other: Standard Care Diet — The standard care diet provides macronutrients within standard amounts (40% carbohydrate, 20% protein, 40% fat) at all meals and snacks per day.
  Arms: Standard Care Diet

SUMMARY:
Gestational diabetes (GDM) is a condition of high blood glucose (or "blood sugar") during pregnancy. GDM can cause harmful short-term and long-term health effects for mom and baby. Diet therapy is an effective way to achieve normal blood glucose for women with GDM, but the best diet is unknown. Diet strategies that improve blood glucose in GDM and that patients can follow are needed for better clinical care. In studies of non-pregnant individuals with diabetes, eating a high fat/protein breakfast as the only dietary change was enough to improve glucose control. Because highest blood glucose readings in GDM usually occur after breakfast, a high fat/protein breakfast could also improve glucose control in GDM. In this study, two dietary strategies for improving blood glucose will be compared. Ten women newly diagnosed with GDM (<30 weeks in pregnancy) will be enrolled in a 12-day cross-over controlled feeding study with a high fat/protein breakfast, which is named a 'Macro-Optimized Diet' (MOD) or standard care diet (SC). In other words, subjects will have all food provided to them, and they will consume each diet for a few days while researchers monitor their blood glucose. Most nutrition aspects of the two diets will be similar, but the MOD diet will vary the timing of eating carbohydrate, protein, and fat to achieve fewer carbs at breakfast. After the 12-day controlled feeding period, participants will continue one of the study diets (as randomized) until delivery. During this time, research team dietitians will provide personalized nutrition education to support GDM self-management. The study will evaluate whether the diet is acceptable to women with GDM and their clinic providers. Data to be collected include blood glucose data, patient and provider feedback on diet acceptability, weight gain, the number of participants who are prescribed blood glucose control medications, and infant weight. These data will be used to evaluate trends pointing to whether one diet is more effective.

DETAILED DESCRIPTION:
Study Objectives: This research proposes to evaluate the feasibility of the proposed two-phased study: 1) compare two diet strategies to management of Gestational Diabetes Mellitus via a 12-day randomized cross-over feeding study, and 2) support patient self-management of assigned diet for remainder of pregnancy with clinical management team.

Study Type and Design:

1. Type/Design: Single-center, randomized controlled cross-over feeding study
2. Intervention and Control Procedures:

   1. Women between the ages of 18-40 years attending the University of Kansas Medical Center's high-risk clinic with a positive GDM diagnosis will be recruited.
   2. Randomization will occur after consent and will determine: 1) the first study diet for the 12-day cross-over controlled feeding, and 2) the 2nd study diet for the 12- day cross-over controlled feeding, which will be continued as the study diet for the remainder of pregnancy.
   3. All food will be provided to participants during the 12-day controlled feeding period.

      Consented women will report to the Clinical Research Center (CRC) on day 1 to collect venous blood samples and receive 2 days of wash-out diet. Participants will return on day 3 fasting for placement of the continuous glucose monitoring system (CGMS) and to collect 3 days of the first randomly assigned study diet (MOD or SC). On day 6, participants will return to the CRC fasting, provide a blood sample, and remove the CGMS. They will be served a breakfast for the first study diet, and hourly blood samples will be collected for 5 hours. After all blood samples have been collected, participants will receive wash-out diet meals/snacks through day 8.

      The same protocol will be repeated for days 9-12 for the alternative study diet (MOD or SC).
   4. At the completion of the 12-day cross-over controlled feeding study, participants will continue with the SC or MOD study diets (the last diet followed after randomization) to implement with registered dietitian (RD) support for the remainder of the pregnancy. Food will not be provided by the study team for this portion of the study. Standard care guidelines for dietetics practice in GDM recommend three visits with a registered dietitian. These visits will take place as as two face-to-face and two telephone encounters.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages 18-40 years old
* A positive GDM diagnosis at 24-28 weeks gestation
* GDM management by diet alone
* willing to consume food provided in the study
* English speaking

Exclusion Criteria:

* multiple gestation
* hypertriglyceridemia (fasting TG >400 mg/dL)
* suspected overt diabetes (previous A1c≥6.5)
* smoker
* fasting glucose >110mg/dL
* overt cognitive impairment
* presence of risk factors for placental insufficiency or growth restriction (e.g.

hypertension, renal disease, history of preeclampsia, use of β-blockers)

* history of preterm birth
* other major medical disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Diet Satisfaction | 18 months
  Diet satisfaction will be measured by the Diet Satisfaction Questionnaire (James et al, 2018), a 28-item validated survey that measures diet satisfaction on 7 scales (healthy lifestyle, convenience, cost, family dynamics, preoccupation with food, negative aspects, and planning and preparation). Item statements are rated by participants on a 5-point Likert scale. Acceptability of both diets will be evaluated by degree of agreement with survey items using means +/- standard deviations for 7 subscales of diet satisfaction.
Adherence to the study diet | 18 months
  Adherence to the study diet will be measured during both phases of the study. During the controlled feeding portion of the study, participants will log their % consumption of all meals and snacks and return logs to the research team. For the self-monitored phase, three multiple pass 24 hour dietary recalls will be collected by trained staff.
  Macronutrient analysis of 24 hour recalls will be evaluated by eating occasion to determine diet adherence. Participants will also keep daily logs for food intake at breakfast. Logs will be sent weekly to the study team electronically. Adherence will be calculated as number of days meeting macronutrient goals at breakfast for both 24 hr recalls and logs. Participants will be considered adherent if meeting goal at least 75% of the time.

SECONDARY OUTCOMES:
Glucose Incremental area under the curve (iAUC) | 12 months
  iAUC measures glycemic excursions after meals and is calculated from glucose measurements using the trapezoid method38
Prescription rates | 18 months
  Frequency of prescription of glucose lowering medication after study enrollment
Gestational weight gain | 18 months
  Body weight gained between study enrollment and delivery.
Infant weight | 18 months
  Infant weight at birth in grams

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Gibbs, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No